CLINICAL TRIAL: NCT06455371
Title: Patient-centered Decision Support Tool for Levothyroxine Dosage
Brief Title: Patient-centered Dosage of Levothyroxine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: SINTEF Health Research (Other); Helseapps (Unknown); Norinnova (Unknown); Helse Nord (Industry)
Responsible Party: Principal Investigator, Vegard Brun, Consultant physician and associate professor, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 547311
Record Dates: First submitted 2024-01-10; First posted 2024-06-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-12

CONDITIONS: Hypothyroidism; Thyroid Cancer; Thyroid
Keywords: Decision support tool; Patient-centered dosage; thyroidectomy; levothyroxine
MeSH Terms: conditions — Hypothyroidism; Thyroid Neoplasms; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention): Current clinical practise. Levothyroxine dose is calculated based on weight and adjusted according to TSH-level at 6-8 week intervals until biochemical target is reached
- DST 1 (Experimental): Levothyroxine dose is calculated using the current version of the decision support tool based on 4 blood samples.
  Interventions: Other: Decision support tool
- DST 2 (Experimental): Levothyroxine dose is calculated using an improved mathematical model in the decision support tool based on 4 blood samples.
  Interventions: Other: Decision support tool
- DST 3 (Experimental): Levothyroxine dose is calculated using an improved mathematical model in the decision support tool based on 2 blood samples.
  Interventions: Other: Decision support tool

INTERVENTIONS:
Other: Decision support tool — Patients in the intervention groups are given the option to use the decision support tool when adjusting the levothyroxine dose after total thyroidectomy. Levothyroxine therapy is not a part of the intervention, as all patients receive this therapy regardless of study participation.
  Arms: DST 1; DST 2; DST 3

SUMMARY:
Levothyroxine is the most used thyroid hormone replacement when the thyroid gland is failing. Because dosage adjustment normally takes several months, the investigators have developed a decision support tool (DST) that predicts optimal dosage based on repeated blood samples the first 2 weeks after initiation of therapy. In this randomized study the investigators will include patients that start levothyroxine therapy after total thyroidectomy. The use of DST to advice the physician about an early dosage adjustment will be compared with common clinical practice, that is dosage adjustment every 2 months. The effect of DST use will be assessed by studying the possible relationship between fast optimal dose adjustment, patient reported outcome measures, and ability to work.

ELIGIBILITY:
Inclusion Criteria:

* Total or completion thyroidectomy for differentiated thyroid cancer og benign thyroid nodules at Norwegian hospitals

Exclusion Criteria:

* Anaplastic thyroid cancer, thyroid cancer with distant metastasis, graves disease, toxic nodules, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients at biochemical target | Outcome is measured at 8 weeks, 6 months and 12 months post surgery
  Number of patients at biochemical target. Biochemical target is TSH (thyroid stimulating hormone) 0,5-2,0 mIE/L for patients on substitution therapy and 0,1-0,5 mIE/L for patients on suppression therapy

SECONDARY OUTCOMES:
Time to biochemical target | Measured at 18 months after surgery
  Time to biochemical target is reached measured in days. Day 0 is day of surgery
Distance from biochemical target | Measured at 8 weeks post surgery
  Distance measured in TSH units.
Patient reported outcome - ThyPRO39 questionnaire | Measured at 2 weeks before surgery, 2 months after surgery and 6 months after surgery surgery
  Patient reported outcomes measured by the validated questionnaire ThyPRO39. The ThyPRO39 questionnaire consist of 12 scales that covers physical symptoms (goiter, eye symptoms, hypo- and hyperthyroid symptoms), cosmetic appearance, physical, mental and social well-being and function. Each item is rated on a 0-4 scale from 0 = no symptoms/problems to 4 = Severe symptoms/problems. The average score of items in a scale is divided by four and multiplied by 100 to yield thirteen 0-100 scales, with higher scores indicating worse health status.
  The questionnaire will be distributed three times during the study. The first measurement will be two weeks before surgery and represent the baseline. The questionnaire is distributed again at 2 months and 6 months after surgery and changes from baseline will be measured and compared between groups.
Patient reported outcome - RAND-36 questionnaire | Measured at 2 weeks before surgery, 2 months after surgery and 6 months after surgery surgery
  Rand-36 is the Norwegian translation of the SF-36 version 1.2. The questionnaire consists of 36 items, grouped into eight multi-item scales that measure physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health. The scores can also be summarized into two summary scores for overall physical and mental health. Items scores will be transformed to 0-100 point scales (0=worst, 100=best) using the SF-36 scoring algorithm
  The questionnaire will be distributed three times during the study. The first measurement will be two weeks before surgery and represent the baseline. The questionnaire is distributed again at 2 months and 6 months after surgery and changes from baseline will be measured and compared between groups.
Abscence from work | Measured at18 months after surgery
  Days with sick-leave from work the first year after surgery. Data collected from the Norwegian national sick-leave registry

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brun VH, Eriksen AH, Selseth R, Johansson K, Vik R, Davidsen B, Kaut M, Hellemo L. Patient-Tailored Levothyroxine Dosage with Pharmacokinetic/Pharmacodynamic Modeling: A Novel Approach After Total Thyroidectomy. Thyroid. 2021 Sep;31(9):1297-1304. doi: 10.1089/thy.2021.0125. Epub 2021 Jun 22. PMID 33980057